CLINICAL TRIAL: NCT01166581
Title: Evaluation of Breast Magnetic Resonance Imaging (MRI) Impact on Mastectomy Rate at Summa Akron City Hospital
Brief Title: Impact of Breast Magnetic Resonance Imaging (MRI) on Mastectomy Rates
Status: Terminated | Type: Observational
Why Stopped: Not enough data collected to work with
Sponsor: Summa Health System (Other)
Responsible Party: Sponsor
Other Study IDs: Doncals Breast MRI study
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Early Stage Breast Cancer
Keywords: early stage breast cancer; preoperative breast MRI; mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of this study is to determine if preoperative breast MRI findings resulted in more extensive surgery, i.e., mastectomy than breast conserving surgery, i.e., lumpectomy in early stage breast cancers at Summa Akron City Hospital. Early stage breast cancer is defined as breast tumor size less than 5 cm.

The objectives are to:

* Review early stage breast cancer patient cases treated at Summa Akron City Hospital between 2006 and 2009 to evaluate clinical and pathological staging
* Determine the results of preoperative breast MRI and the impact on type of surgery performed
* Evaluate the decision to have mastectomy rather than lumpectomy, i.e., physician or patient decision and if this decision was based on breast MRI findings

DETAILED DESCRIPTION:
Early stage breast cancer cases between 2006 and 2009 will be identified by the Summa Akron City Hospital cancer registry. The cases will be reviewed and abstracted. The abstracted data will include results of physical breast examinations, mammograms, sonograms, breast MRI reports, biopsy procedure notes and pathology reports to illustrate the clinical stage. Definitive surgical pathology reports will be included in the abstracted data to demonstrate the final pathologic stage of the breast cancer.

A database will be developed to capture the abstracted data. Outcomes will be determined based on final pathology reports.

ELIGIBILITY:
Inclusion Criteria:

* early stage breast cancer between 2006-2009
* preoperative MRI

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: early stage breast cancer cases between 2006-2009
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to determine if preoperative breast MRI findings resulted in more extensive surgery than breast conserving surgery in early stage breast cancers at Summa Akron City Hospital. | from 2006-2009
  Review early stage breast cancer patient cases treated at Summa Akron City Hospital between 2006 and 2009 to evaluate clinical and pathological staging
  Determine the results of preoperative breast MRI and the impact on type of surgery performed
  Correlate the breast MRI findings with the final pathology results to determine if the breast MRI clinically upstaged the cancer.

SECONDARY OUTCOMES:
Correlate the breast MRI findings with the final pathology results to determine if the breast MRI clinically upstaged the cancer | 2006-2009

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Doncals, MD, Principal Investigator — Summa Health System
Locations (1):
- Summa Akron City Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Del Frate C, Borghese L, Cedolini C, Bestagno A, Puglisi F, Isola M, Soldano F, Bazzocchi M. Role of pre-surgical breast MRI in the management of invasive breast carcinoma. Breast. 2007 Oct;16(5):469-81. doi: 10.1016/j.breast.2007.02.004. Epub 2007 Apr 12. PMID 17433681
- [Background] Ciocchetti JM, Joy N, Staller S, Warmack J, Mann A, Moore JT, Davis-Merritt DK. The effect of magnetic resonance imaging in the workup of breast cancer. Am J Surg. 2009 Dec;198(6):824-8. doi: 10.1016/j.amjsurg.2009.05.029. PMID 19969136